CLINICAL TRIAL: NCT02633046
Title: Treatment of Proteinuria Due to Treatment Resistant or Treatment Intolerant Idiopathic Focal Segmental Glomerulosclerosis: A Prospective Study of Acthar (PODOCYTE)
Brief Title: Acthar for Treatment-Resistant or Treatment-Intolerant Proteinuria
Acronym: PODOCYTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mallinckrodt ARD LLC (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNK14224049
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Idiopathic Focal Segmental Glomerulosclerosis
Keywords: FSGS; primary FSGS; idiopathic FSGS
MeSH Terms: interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acthar Gel (Other): Acthar Gel, 1 mL (80 U) by subcutaneous injection (SC) 3x/week will be administered to all participants from Week 0 to 50. Tapering of dose to 1 mL SC 2x/week will be allowed for safety and/ tolerability issues. Once the dose is tapered to 1 mL SC 2x/week it must remain at this level. Participants unable to tolerate 1 mL SC 2x/week will be discontinued. All participants will have an End of Study/Early Termination Visit 4 weeks after discontinuing Investigational Medicinal Product (IMP).
  Interventions: Drug: Acthar Gel

INTERVENTIONS:
Drug: Acthar Gel — Acthar Gel 80 U/mL solution for subcutaneous injection
  Other Names: Acthar

SUMMARY:
Focal segmental glomerulosclerosis (FSGS) is a condition that harms the kidney "filters" that remove waste from the blood. Proteins are supposed to stay in the blood. Damaged "filters" let protein get into the kidney.

FSGS is a serious condition that can lead to kidney failure. The only treatment for kidney failure is dialysis or kidney transplant.

Proteinuria means too much protein came through the kidneys into the urine.

If the doctor cannot figure out what is causing the problem, it is primary (idiopathic) FSGS. This kind of FSGS is very hard to treat.

This study will test Acthar in patients with this condition who have not responded to other treatments. It primarily investigates how well the therapy is tolerated by the patients and how well they respond to this treatment.

ELIGIBILITY:
Inclusion Criteria

Potential participants must meet the following summary criteria for inclusion in the study:

* Is male or non-pregnant, non-lactating female
* Has primary FSGS, is nephrotic and did not achieve at least partial proteinuria response with prior therapy
* Has been treated with an angiotensin converting enzyme inhibitor or receptor blocker (or have documented intolerance), for at least 4 weeks before screening
* Has blood pressure no higher than 150/90 mmHg
* Meets all other inclusion criteria detailed in the protocol

Exclusion Criteria

Potential participants will not be eligible for the the study if they meet the following summary criteria:

* Has hepatitis B or C, tuberculosis, or other contraindication listed on the United States (US) Prescribing Information for Acthar
* Has Type 1 or Type 2 diabetes mellitus or any clinically significant infection
* Has received specific treatments at exclusionary time points per protocol
* Has been involved in a therapeutic drug/device trial (other than for FSGS) within 4 weeks before screening
* Meets any other exclusion criteria detailed in the protocol
* Has any other condition that might, per protocol or in the opinion of the investigator, compromise:

  1. the safety and well-being of the participant or their offspring
  2. the safety of study staff
  3. analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (47):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - AKDHC Medical Research Services, LLC, Tucson, Arizona
  - California Institute of Renal Research, Chula Vista, California
  - Stanford University, Stanford, California
  - VERITAS Research Corp, Miami Lakes, Florida
  - Genesis Clinical Research Corp, Tampa, Florida
  - GA Nephrology, Lawrenceville, Georgia
  - NANI Research, Hinsdale, Illinois
  - University of Louisville Research Foundation, Inc., Louisville, Kentucky
  - Ochsner Clinic Foundation, Baton Rouge, Baton Rouge, Louisiana
  - NKDHC Medical Research Services, LLC, Las Vegas, Nevada
  - Icahn School of Medicine-Mt. Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Metrolina Nephrology Associates, Charlotte, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - University of Cincinnati Physicians Company, LLC, Cincinnati, Ohio
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Tech University Health Science Center, Amarillo, Texas
  - Texas Kidney Institute (Neprhotex Research Group), Dallas, Texas
  - University of Wisconsin Wisconsin Dialysis Institute, Madison, Wisconsin
- Argentina (3):
  - Centro de Salud Renal Junín SRL, Junín, Buenos Aires
  - Centro de Investigaciones Médicas, Mar del Plata, Buenos Aires
  - Sanatorio Allende, Córdoba
- Australia (7):
  - Renal Research Group, Gosford, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospita, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Launceston Hospital, Launceston, Tasmania
  - The Alfred Hospital, Melbourne, Victoria
  - Sunshine Hopital - Western Health, St Albans, Victoria
- Chile (2):
  - Hospital Dr. Hernán Henríquez Aravena, Temuco, Región de la Araucanía
  - Clinica Davila, Santiago, RM
- Mexico (2):
  - Investigación Nefrológica SC, Cuernavaca, Morelos
  - Hospital y Clínica OCA S.A de C.V, Monterrey, Nuevo León
- Peru (4):
  - Hospital Nacional Cayetano Heredia, San Martín de Porres, Lima region
  - Hospital Nacional Alberto Sabogal, Lima
  - Hospital Nacional Arzobispo Loayza, Lima
  - Hospital Nacional Hospital Maria Auxiliadora, Lima Lima
- Turkey (Türkiye) (8):
  - Şişli Etfal Hamidiye Training and Research Hospital, Istanbul, Sisli
  - İstanbul University Faculty of Medicine, Istanbul, Topkapi
  - Ankara NumuneTraining and Research Hospital, Ankara
  - Ankara Training and Research Hospital, Ankara
  - İstanbul University Faculty of Medicine, Istanbul
  - Kocaeli University Faculty of Medicine, Kocaeli
  - Marmara University Faculty of Medicine, Maltepe
  - Mersin University Faculty of Medicine, Mersin

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT02633046) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

REFERENCES:
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multiple locations enrolled participants in Argentina (3), Australia (5), Chile (4), Mexico (5), Peru (8), Turkey (13), and the United States (25).
Groups:
- Acthar Gel: All participants receive open-label treatment with Acthar Gel per protocol regimen:
  Acthar Gel, 1 mL (80 U) by subcutaneous injection (SC) 3x/week will be administered to all participants from Week 0 to 50. Tapering of dose to 1 mL SC 2x/week will be allowed for safety and/ tolerability issues. Once the dose is tapered to 1 mL SC 2x/week it must remain at this level. Participants unable to tolerate 1 mL SC 2x/week will be discontinued. All participants will have an End of Study/Early Termination Visit 4 weeks after discontinuing Investigational Medicinal Product.
Period: Overall Study
Arm/Group | Acthar Gel
Started | 63
Safety Population | 63
Completed | 36
Not Completed | 27
Not completed — Adverse Event | 8
Not completed — Physician Decision | 7
Not completed — Withdrawal by Subject | 8
Not completed — Increased proteinuria | 2
Not completed — Participant decided not to continue with open label extension | 1
Not completed — Mutual decision patient and physician | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set, defined as all participants allocated to study treatment
Groups:
- Acthar Gel: All participants receive open-label treatment with Acthar Gel per protocol regimen
Arm/Group | Acthar Gel
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (13.54)
Age, Customized [Count of Participants; unit: Participants]
  18-25 years of age | 16
  26-45 years of age | 29
  46-65 years of age | 17
  greater than 65 years of age | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants who selected multiple races or identified themselves as mixed-race are included in the Unknown category.
  Participants
    American Indian or Alaska Native | 2
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 4
    White | 48
    More than one race | 0
    Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  Argentina | 3
  Turkey | 13
  United States | 25
  Mexico | 5
  Australia | 5
  Chile | 4
  Peru | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Clinically significant changes in laboratory or physical examination findings are counted as adverse events. Descriptive statistics are collected for participants with:
  1. death for any reason (all cause mortality)
  2. treatment emergent serious adverse events (TESAEs)
  3. any non-serious treatment emergent adverse events (TEAEs)
Time Frame: within 56 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar Gel
Number analyzed (Participants) | 63
Participants
  Deaths | 0
  Serious TEAEs | 11
  Non-serious TEAEs | 60

ADVERSE EVENTS:
Time Frame: within 56 weeks
Description: Treatment emergent adverse events are recorded.
Arm/Group | Acthar Gel
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 11/63
Other Adverse Events (participants affected / at risk) | 50/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acthar Gel (N=63)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Oedema (General disorders) | 1 (2)
Pyrexia (General disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (2)
Blood creatinine increased (Investigations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acthar Gel (N=63)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 5 (6)
Injection site bruising (General disorders) | 5 (5)
Oedema (General disorders) | 10 (13)
Oedema peripheral (General disorders) | 5 (7)
Nasopharyngitis (Infections and infestations) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 14 (15)
Weight increased (Investigations) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Headache (Nervous system disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 9 (9)
Hypertension (Vascular disorders) | 10 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT02633046/Prot_SAP_000.pdf